CLINICAL TRIAL: NCT05679635
Title: Evaluation of Tracheal Pressure During Continuous Positive Airway Pressure Ventilation - a Prospective, Clinical Trial
Brief Title: Evaluation of Tracheal Pressure During CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1224/2022
Record Dates: First submitted 2022-11-28; First posted 2023-01-11 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Continuous Positive Airway Pressure; CPAP Ventilation
Keywords: tracheal pressure; airway pressure

STUDY DESIGN:
Intervention Model Description: prospective, open, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Other): In intubated patients during CPAP ventilation, a conventional tube adapter (CTA, Ventinova Medical B.V., Eindhoven, The Netherlands) will be connected to the tracheal tube for tracheal pressure measurement. Tracheal pressure measurements will be recorded directly from the respirator Evone (Ventinova Medical B.V., Eindhoven, The Netherlands) three times, as well as the corresponding airway pressure values from the Evita Infinity V500 respirator (Dräger Medical, Lübeck, Germany).
  Study related time points:
  T1: 10 minutes after insertion of the conventional tube adapter during CPAP without ventilator support T2: 10 minutes after T1 during CPAP with activated automatic tube compensation (ATC) T3: 10 minutes after T2 during CPAP with assisted spontaneous breathing (ASB) of 4 cmH2O
  Interventions: Device: Evone; Device: Evita Infinity V500

INTERVENTIONS:
Device: Evone — The conventional tube adapter (CTA) from the Evone ventilator (Ventinova Medical B.V., Eindhoven, The Netherlands), equipped with an tracheal pressure measurement catheter will be connected to the tracheal tube of intubated intensive care unit patients. Subsequently tracheal pressure values will be displayed and recorded from the ventilator.
Device: Evita Infinity V500 — Displayed airway pressure values will be directly recorded from the Evita Infinity V500 ventilator (Dräger Medical, Lübeck, Germany)

SUMMARY:
This trial evaluates tracheal pressure values in intubated intensive care unit patients during continuous positive airway pressure without any ventilatory support, automatic tube compensation and assisted spontaneous breathing.

DETAILED DESCRIPTION:
Aim of this trial is to investigate if there are any significant differences between airway and tracheal pressure values during continuous positive airway pressure (CPAP) ventilation. For this purpose, a tracheal pressure measurement catheter is inserted into the tracheal tube and the obtained values are compared with the corresponding airway pressure measured on the ventilator. To further evaluate the impact of mild respiratory support automatic tube compensation and assisted spontaneous breathing with 4 cmH2O will be applied and measured pressure values compared as well.

We hypothesize that tracheal pressure will be significantly lower than airway pressure values during inspiration, which represents the primary outcome measure. Secondary outcome parameters include comparison of expiratory and mean pressure values of airway and tracheal pressure. Additionally, effects of mild respiratory support will be evaluated as well.

Measurement of inspiratory tracheal pressure might allow to calculate the pressure drop between the airway pressure at the Y-piece of the ventilator and the pressure at the trachea. Currently it is not known, if this pressure drop is significant during CPAP, which represents the rationale to perform this pilot study. In a second step it would be possible to determine if the recorded pressure drop can be used as a surrogate parameter for the respiratory drive in terms of a risk assessment for the development of patient self-inflected lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years
* Intubated patient during CPAP without pressure support
* Informed consent

Exclusion Criteria:

* Female subjects known to be pregnant
* Known participation in another clinical trial
* Critical pulmonary state (paO2/FiO2 ratio <100)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
inspiratory tracheal pressure | 10 minutes after insertion of the tracheal pressure measurement catheter
  The lowest tracheal pressure value, representing the highest inspiratory effort, will be recorded from the ventilator

SECONDARY OUTCOMES:
peak tracheal pressure | 10 minutes after insertion of the tracheal pressure measurement catheter
  The highest tracheal pressure value will be recorded
mean tracheal pressure | 10 minutes after insertion of the tracheal pressure measurement catheter
  The mean tracheal pressure value will be calculated
inspiratory tracheal pressure during automatic tube compensation (ATC) | 10 minutes after adding ATC
  Effect of a mild respiratory support in terms of automatic tube compensation (ATC) on inspiratory tracheal pressure will be evaluated.
inspiratory tracheal pressure during assisted spontaneous breathing (ASB) | 10 minutes after adding ASB
  Effect of a mild respiratory support in terms of assisted spontaneous breathing (ASB) with 4 cmH2O on inspiratory tracheal pressure will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Rugg, MD, Principal Investigator — Medical University of Innsbruck, Department of Anesthesiology and Intensive Care Medicine
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No